CLINICAL TRIAL: NCT02908646
Title: Comparing of Computed Tomography Guided Microcoil Localization and Hook Wire Localization for Pulmonary Small Nodules and Ground-glass Opacity Prior to Thoracoscopic Resection
Brief Title: Comparing of Microcoil Localization and Hook Wire Localization for Resectable Pulmonary Small Nodules
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Pro, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014PHB113
Record Dates: First submitted 2016-09-17; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- microcoil (Experimental): patients who plan for microcoil localization
  Interventions: Procedure: microcoil localization
- hookwire (Placebo Comparator): patients who plan for hookwire localization
  Interventions: Procedure: hookwire localization

INTERVENTIONS:
Procedure: microcoil localization — CT-guided localization by placing a microcoil into the lung parenchyma
  Arms: microcoil
Procedure: hookwire localization — CT-guided localization by placing a hookwire into the lung parenchyma
  Arms: hookwire

SUMMARY:
Both of microcoil localization and hookwire localization have been proved as good preoperative CT(computed tomography)-guided techniques to guide VATS resection for the diagnosis of small peripheral pulmonary nodules technique to guide VATS resection for the diagnosis of small peripheral pulmonary nodules. The objective of this study is to determine if microcoil localization for pulmonary nodules can be safer than hookwire localization

DETAILED DESCRIPTION:
Both of microcoil localization and hookwire localization have been proved as good preoperative CT-guided techniques to guide VATS resection for the diagnosis of small peripheral pulmonary nodules technique to guide VATS(video assisted thoracoscopic surgery) resection for the diagnosis of small peripheral pulmonary nodules. Compared with the commonly used hook wire, the platinum microcoil can be retained in the patients'body and the configuration of which had an effect in reducing the severity of complications. The fibered microcoil may promote blood coagulation of the surrounding lung tissues, block the needle pathway, and decrease the severity of pneumothorax and bleeding caused by the puncture needle, which has been proven in animal experiments. The objective of this study is to determine if microcoil localization for pulmonary nodules can be safer than hookwire localization

ELIGIBILITY:
Inclusion Criteria:

* solid nodules with a diameter ≤1 cm and distance to visceral pleura ≥0.5 cm, -ground-glass nodules,
* part-solid ground-glass nodules, with a solid portion ≤1 cm and distance to the visceral pleura ≥1 cm.
* peripheral nodules amenable to thoracoscopic wedge excision of the nodules.

Exclusion Criteria:

* Patients combined with pneumothorax.
* Patients combined with pleural effusion.
* Patients with history of hemoptysis.
* Patients with medical condition that the radiologist and surgeon disagree for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
complications after CT-guided localization | 1 years
  any complication occured after CT-guided localization

SECONDARY OUTCOMES:
major complications after CT-guided localization | 1 years
  major complication refers to complication that need to be interfered before surgery
success of the intervention of localization | 1 year
  success of the intervention of CT guided localization by microcoil or hookwire
success of the localization by thoracoscopic surgery | 1 year
  success of the localization by thoracoscopic surgery under the guide of the planted microcoil or hookwire

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhao, MD, Principal Investigator — Department of Thoracic Surgery, Center for Mini-invasive Thoracic Surgery, People's Hospital, Peking University
Locations (1):
- Peking university people's hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
no plan to make individual participant data (IPD) available